CLINICAL TRIAL: NCT04318639
Title: The Combination of Donepezil and Cognitive Training for Treating Alcohol Use Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Morris Bell, Senior Research Career Scientist, VA Connecticut Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MB0020
Record Dates: First submitted 2020-03-16; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Alcohol Use Disorder; Mild Cognitive Impairment
Keywords: Alcohol Use Disorder; Mild Cognitive Impairment; Cognitive Remediation Therapy; Donepezil; Recovery
MeSH Terms: conditions — Alcoholism; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Open-label single group design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Donepazil+CRT (Experimental): Donepazil+CRT
  Interventions: Combination Product: Donepazil

INTERVENTIONS:
Combination Product: Donepazil — Donepezil: Subjects will take 5 mg/day of donepezil in the evening for first 4 weeks, then 10 mg/day of donepezil in the evening until week 13.
  Cognitive remediation therapy (CRT): This study employs a computerized program (BrainHQ) for cognitive enhancement. Participants use their program for one hour per session, up to five sessions per week, over 13 weeks (maximum of 65 sessions). They may training on site or at another quiet location of their choice.
  Other Names: Cognitive Remediation Therapy

SUMMARY:
This is an open label feasibility trial to learn whether the combination of donepezil and cognitive remediation therapy (Donepezil + CRT) may improve neurocognitive functioning and decreasing alcohol use in Veterans with alcohol use disorder who have mild cognitive impairment (AUD-MCI). The study will determine the acceptability and adherence to treatment and preliminary evidence for efficacy. The study will recruit 15 newly recovering Veterans individuals with AUD-MCI for a 13-week, open-label, single-arm pilot study with sobriety and cognitive assessments at baseline and at 13-week follow-up.

DETAILED DESCRIPTION:
Donepezil is FDA approved for treatment of dementia and recent animal studies have suggested that it may reduce craving in rat models of alcohol use disorder. Investigators' previous studies of cognitive remediation therapy (CRT) with work therapy have shown efficacy with newly recovering Veterans with AUD compared with work therapy alone. The current study combines Donepezil and CRT in an open-label trial to learn whether the combination of Donepezil + CRT may improve neurocognitive functioning and decrease alcohol use in Veterans with alcohol use disorder who have mild cognitive impairment (AUD-MCI). The study will determine the acceptability and adherence to treatment and provide preliminary evidence for efficacy. The study will recruit 15 newly recovering Veterans individuals with AUD-MCI for a 13-week, open-label, single-arm pilot study with sobriety and cognitive assessments at baseline and at 13-week follow-up. Primary outcome variables will be a Clinical Global Index of AUD recovery and a Global Cognitive Composite of MCI related neurocognitive assessment.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 21-80 years of age
* Fluency in English and a 6th grade or higher reading level
* Meets DSM-V criteria for a current Alcohol Use Disorder
* Referred for the study within 30 days of detoxification or last substance use according to medical records
* Willingness to attend follow-up assessments at 13 weeks
* Willingness to submit to Breathalyzer screenings and Urine Toxicology screenings.
* Meets MCI criteria with greater than 1.5 SD below pre-morbid IQ estimate or 1.5 SD below standard norms on at least 1 key neurocognitive MCI related variable (Learning and Memory, Delayed Recall, Executive Function, Working Memory).

Exclusion Criteria:

* Lifetime diagnosis of a psychotic disorder, not induced by drug use.
* Current prescribed treatment of opioids or benzodiazepines, which may affect new learning Involvement in a legal case that may lead to incarceration during study period
* Residential plans that would interfere with participation
* Medical illness that may significantly compromise cognition (e.g. Parkinson's, Alzheimer's, Huntington's Chorea, Moderate or greater TBI).
* An uncorrected sensory impairment (hearing or sight) that would seriously interfere with cognitive training.
* Pre-morbid IQ estimate below 70.
* Unstable housing or lack of commitment to staying within a geographic area that would make follow-up possible.
* Unwillingness to provide contact information of someone who can help study staff contact the participant in the event that study staff are unable to maintain contact directly.
* Allergy to Donepezil.
* Unstable cardiovascular disease or unstable medical condition-clinically determined by a physician.
* Imminent suicidal or homicidal risk.
* Pregnant or nursing women, positive pregnancy test, or inadequate birth control methods in women of childbearing potential.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical Global Index of AUD recovery | 13 weeks
  7-point likert scale of recovery
Global Composite T-Score of MCI related neurocognitive measures. | 13-week
  Measures of Learning and memory, delayed recall, working memory and executive. Higher scores indicate better functioning

OTHER OUTCOMES:
Feasibility and Acceptability of Interventions | 13 weeks
  Adverse events
Adherence to Donepezil | 13 weeks
  Percentage of Donepezil compliance based on weekly pill counts
Adherence to CRT | 13 weeks
  Percentage of training sessions completed out of 65 possible sessions

CONTACTS AND LOCATIONS:
Overall Officials: Morris Bell, Principal Investigator — VA Connecticut Healthcare System
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Only those already identified in HIPAA

REFERENCES:
- [Result] Mulholland PJ, Teppen TL, Miller KM, Sexton HG, Pandey SC, Swartzwelder HS. Donepezil Reverses Dendritic Spine Morphology Adaptations and Fmr1 Epigenetic Modifications in Hippocampus of Adult Rats After Adolescent Alcohol Exposure. Alcohol Clin Exp Res. 2018 Apr;42(4):706-717. doi: 10.1111/acer.13599. Epub 2018 Feb 15. PMID 29336496
- [Result] Bell MD, Laws H, Pittman B, Johannesen JK. Comparison of focused cognitive training and portable "brain-games" on functional outcomes for vocational rehabilitation participants. Sci Rep. 2018 Jan 29;8(1):1779. doi: 10.1038/s41598-018-20094-w. PMID 29379114